CLINICAL TRIAL: NCT06726083
Title: Improving Dietary Quality and Social Engagement Through a Virtual Nutrition and Teaching Kitchen Intervention Among Older Veterans With Impaired Mobility
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E5306-R
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Impaired Mobility
Keywords: diet quality
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with an intervention group compared to a control group
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to study participant group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nutrition Intervention (Experimental): Weekly virtual live group sessions led by a trained study team member will be held twice weekly for 1 hour/week over 12 weeks using a HIPAA compliant online platform. The first class of each week will include the teaching kitchen cooking demonstration (~30 min) and the remainder of the class will focus on dietary education. The second class each week will provide an opportunity for group discussion to have Veterans share to their peers about how they used the weekly produce
  Interventions: Behavioral: Nutrition Intervention
- Contact Control (Active Comparator): Weekly virtual live group health education sessions led by staff will be held for two hours/week over 12 weeks. We will enroll up to 15 participants into each virtual class cohort and run multiple different group sessions for a total sample size of 90 participants. The content follows the LIFE study structured successful aging health education curriculum80,81 which was designed to increase self-efficacy and empower older Veterans to take control of their own healthcare. Topics focus on a broad range of healthy aging, such as importance of sleep, safe travel, goal setting, self-care, and common comorbidities
  Interventions: Behavioral: Contact Control

INTERVENTIONS:
Behavioral: Nutrition Intervention — Weekly virtual live group sessions led by a trained study team member will be held twice weekly for 1 hour/week over 12 weeks using a HIPAA compliant online platform. The first class of each week will include the teaching kitchen cooking demonstration (~30 min) and the remainder of the class will focus on dietary education. The second class each week will provide an opportunity for group discussion to have Veterans share to their peers about how they used the weekly produce
  Arms: Nutrition Intervention
Behavioral: Contact Control — Weekly virtual live group health education sessions led by staff will be held for two hours/week over 12 weeks. We will enroll up to 15 participants into each virtual class cohort and run multiple different group sessions for a total sample size of 90 participants. The content follows the LIFE study structured successful aging health education curriculum80,81 which was designed to increase self-efficacy and empower older Veterans to take control of their own healthcare. Topics focus on a broad range of healthy aging, such as importance of sleep, safe travel, goal setting, self-care, and common comorbidities
  Arms: Contact Control

SUMMARY:
Compared to non-Veterans, Veterans demonstrate an increased risk for obesity and multimorbidity. Thus, interventions to improve overall health are warranted in this population. Healthy diets that include fruits and vegetables are linked to a reduced risk of chronic disease including mobility disability, and are associated with higher muscle mass, strength and physical performance potentially slowing further disability progression later in life. The investigators will determine if a three-month virtual group nutrition intervention paired with produce delivery and virtual teaching kitchen cooking demonstrations tailored for older Veterans with impaired mobility will improve diet, health-related quality of life and muscle strength.

DETAILED DESCRIPTION:
There are >8 million older Veterans (>65 years) in the United States, and nearly half of them self-report having a disability such as impaired mobility that impacts their ability to perform self-care. Among older Veterans with mobility disability, common self-care tasks like food shopping, meal preparation, and cooking are barriers to consuming a healthy diet, resulting in poor dietary intake. Poor dietary intake contributes to chronic disease risk and loss of muscle mass and strength, consequently limiting function and increasing immobility. Teaching older Veterans with impaired mobility how to overcome barriers limiting these diet-related self-care tasks provides an opportunity to significantly impact this group's dietary intake. Lack of social support has also been associated with negative health outcomes and poor nutritional intake; thus, effective, age-friendly intervention strategies to improve dietary quality as a strategy to delay further progression of disability and maintain functional independence among this population are needed.

In this randomized controlled trial, the investigators will determine if a 3-month virtual group nutrition intervention paired with produce delivery and virtual teaching kitchen cooking demonstrations tailored for older Veterans will improve diet and functional mobility. The overarching hypothesis is that virtual group nutrition education classes and cooking demos, personalized to include considerations of this population's physical limitations, age-related taste changes and technological barriers, will result in favorable improvements in dietary quality and functional mobility while promoting social interaction.

Specific Aim 1: determine the impact of the virtual intervention paired with produce delivery and virtual cooking demonstrations on objective measures of diet quality compared to contact control among a diverse sample of older Veterans with impaired mobility. Additionally, the investigators will assess the sustained effects of the program on dietary quality at a 6-month follow-up, 3-months after the virtual intervention ends. If no treatment effects are observed at the end of the 3-month intervention, the investigators will explore reasons why the intervention was ineffective.

Specific Aim 2: determine the impact of the 3-month virtual nutrition intervention on measures of social isolation, health-related quality of life and mental health using validated questionnaires.

Specific Aim 3: determine associations with changes in dietary quality and frailty-related physical function outcomes and body composition among those who benefit from a virtual nutrition education and cooking program.

ELIGIBILITY:
Inclusion Criteria:

* Veterans >65 years with reduced gait speed (gait speed <1.0 m/s) or elevated four square step test
* use of an assistive device who also indicate that they would like to improve their eating habits, defined by response of <3 on a scale of 1 to 5 to the question, 'Do you consider your eating habits to be healthy'

Exclusion Criteria:

* uncontrolled diabetes mellitus or chronic kidney disease
* contraindications to a nutrition intervention including physician prescribed diet (e.g. renal diet)
* dementia (on medical record review or a mini-mental status exam score <24)
* currently participating in a diet or weight loss intervention
* behavior that prevents group interaction

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Diet quality | 3 month and 6 month compared to baseline
  Habitual dietary intake will be assessed using three 24-h recalls via the online Automated Self-Administered 24-hour (ASA24) Dietary Assessment Tool, version (2022), developed by the National Cancer Institute, Bethesda, MD. The dietary recalls will be used to calculate diet quality using the HEI; scores range from 0 to 100; higher scores indicate better adherence to the Dietary Guidelines for Americans.
Social Isolation | 3 month and 6 month compared to baseline
  The Lubben Social Network Scale, is a 12-item scale to assess self-reported social engagement including family and friends (Cronbach's =0.70). The total score is calculated by finding the sum of the all items. The score ranges between 0 and 60, with a higher score indicating more social engagement. The UCLA Loneliness Scale is a 20-item scale to measure subjective feelings of loneliness & social isolation (Cronbach's 0.89<0.94). Using a 4-point rating scale (1= never; 4 = always), participants answer 20 questions, such as "How often do you feel left out?" and "How often do you feel part of a group of friends?" Researchers later reverse-code the positively worded items so that high values mean more loneliness, and then calculate a score for each respondent by averaging their ratings. Both measures are included because they assess complementary but separate constructs

SECONDARY OUTCOMES:
Health-related Quality of Life | 3 month and 6 month compared to baseline
  The PROMIS Global Health (v1.2) consist of 10 items on a 5-pt Likert scale to measure an individual's physical (GPH) and mental health (GMH). The GPH score comprises 4 items on physical health, physical functioning, pain intensity, and fatigue. The GMH score includes 4 items on overall HRQoL, mental health, satisfaction with social activities/relationships, & emotional problems. Higher scores indicate better HRQoL.
Body Composition | 3 month
  Total and regional percentage body fat, absolute fat mass and fat-free mass will be measured using dual energy X-ray absorptiometry (DEXA).
Modified Physical Performance Test (MPPT) | 3 month and 6 month compared to baseline
  The MPPT is a nine-item standardized test used to identify frailty and mobility dysfunction in older individuals. It scores individuals on the time it takes to complete such tasks as donning and doffing a coat, picking a penny from the ground, and ascending the stairs. These scores are then summed out of 36 and scores of less than 32 indicate at least mild frailty.
Functional Gait Assessment (FGA) | 3 month and 6 month compared to baseline
  The FGA is a 10-item clinical gait test that is based on the dynamic gait index (DGI). It tests higher level dynamic gait activities that are part of daily functional mobility such as turning safely and ambulating backwards. Total scores ranging from 0 to 30 and scores below 22 are predictive of future falls.
Falls-Efficacy Scale-International (FES-I) | 3 month and 6 month compared to baseline
  The FES-I is a 16-item self-reported tool that measures fear of falling when completing routine activities such as preparing a meal, going shopping, getting dressed, visiting with friends and family, and reaching up or bending down. The level of concern is measured on a four-point Likert scale (1=not at all concerned to 4=very concerned). It is scored from 16-64 points (high fear of falling >23 points)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Dennis, PhD RD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No